CLINICAL TRIAL: NCT02355288
Title: Left Internal Thoracic Artery Bypass Versus Percutaneous Revascularization in Diabetics:Is Minimally Invasive Left Internal Thoracic Artery Bypass Superior to Percutaneous Revascularization in Diabetic Patients With Isolated LAD Stenosis?
Brief Title: Left Internal Thoracic Artery Bypass Versus Percutaneous Revascularization in Diabetics
Acronym: LIBERTI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient funding available to complete study.
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Principal Investigator, Marc Ruel MD MPH FRCSC, Professor and Chairman, Division of Cardiac Surgery, Ottawa Heart Institute Research Corporation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20130910
Record Dates: First submitted 2014-12-08; First posted 2015-02-04 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-04

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus
Keywords: Coronary Artery Disease; Diabetes Mellitus; Minimally Invasive Cardiac Surgery; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally Invasive Coronary Bypass (Active Comparator): Minimally invasive bypass surgery (MICS CABG) would be conducted to treat the left anterior descending (LAD) artery disease in diabetic patients. This would be a surgical intervention, and differs from the stent procedure arm.
  Interventions: Procedure: Minimally Invasive Coronary Bypass
- Percutenous Coronary Intervention (Active Comparator): Percutaneous coronary intervention (PCI) with drug eluting stents would be used to treat left anterior descending (LAD) artery disease in diabetic patients. This would be an intervention induced by cardiology, and differs from the surgical intervention arm.
  Interventions: Procedure: Percutenous Coronary Intervention

INTERVENTIONS:
Procedure: Minimally Invasive Coronary Bypass — Bypass graft of the Left Anterior Descending (LAD) artery using minimally invasive cardiac surgery. MICS is a bypass surgery done with a small (4-6 cm) incision under the left breast, instead of the usual incision down the middle the chest.
  Arms: Minimally Invasive Coronary Bypass
Procedure: Percutenous Coronary Intervention — Stenting of the Left Anterior Descending (LAD) artery using a drug-eluting stent.
  Arms: Percutenous Coronary Intervention

SUMMARY:
The purpose of this study is to evaluate whether less invasive bypass surgery using the left chest wall artery is more or less effective than inserting a heart stent in patients with diabetes and a blockage of the main artery at the front of the heart. This will be a clinical trial study where the investigators will test the rate of recruitment into the study, as well as the feasibility of allocating each of the 2 treatments.

DETAILED DESCRIPTION:
Purpose/Objectives:

The purpose of this pilot study is to evaluate whether minimally invasive bypass surgery with the left internal thoracic artery (MICS CABG) is more or less effective than percutaneous revascularization with drug eluting stents (PCI/DES) in patients with diabetes and stenosis of the left anterior descending (LAD) artery.

Population:

The investigators will recruit 100 adults with diabetes mellitus (Type 1 or Type 2) and angiographically-confirmed proximal or mid LAD disease, morphologically amenable to either MICS CABG or PCI/DES; outside the context of an acute ST-elevation myocardial infarction, and with indication for revascularization based upon symptoms of worsening angina and/or objective evidence of myocardial ischemia.

Design:

This trial is a multicentre, two-arm, open label, prospective, randomized, pilot trial over a duration of 2.75 years, with 0.75 year of initiation, 1 year of patient recruitment and 2 years of follow-up. Patients who consent will be randomized on a 1:1 basis either to MICS CABG or PCI/DES of the LAD, and followed at 30 days, 6 months, 1 year, 18 months, and 2 years.

Treatment:

Eligible patients will be randomized to receive either MICS CABG or PCI/DES to the LAD. Patients randomized to the PCI/DES arm will receive, at the discretion of the primary physician or interventionalist, the stent of choice at the treating institution, with a recommendation of a everolimus- or zotarolimus-eluting stent.

Primary Endpoint:

The primary endpoint is successfully enrolled, eligible and consenting patients within the first year of enrollment, with success defined as 100 patients or more.

Secondary Endpoints:

All-cause mortality, Myocardial Infarction (MI), stroke and target vessel revascularization (TVR) will be compared for the therapy comparison PCI/DES versus MICS CABG. For these analyses, the survival analysis outlined for the primary analysis will be followed.

Quality of Life (QOL) at 1 month, 6 months, 1 year, 18 months, and 2 year will be compared for the therapy comparison PCI/DES vs. MICS CABG. Patients will be asked to complete the following questionnaires: the EuroQOL (EQ-5D) and Seattle Angina Questionnaire (SAQ).

Statistics:

The main feasibility questions are: "can the investigators enroll a sizable number of patients at a given centre over a 1 year period?", "can the investigators implement and conduct the proposed trial across multiple centres?", and "can the investigators ensure high protocol adherence and follow-up, as well as minimize crossovers?". By enrolling 100 participants across 5 sites over 1 year, and follow them.

For each therapy group, the frequency distribution each of the domains of the EQ5D will be tabulated and the mean, standard deviation, median and interquartile range (IQR) calculated. Therapy groups will be compared on these outcomes using the t-test or the Wilcoxon rank-sum test and 95%CI calculated. Repeated measures ANOVA will compare the two therapy groups on changes in health related QOL over time

Participating Centres:

The investigators have chosen 5 study sites in Canada (3) and in the United States (2). The recruitment goal for each site is to enroll at least 20 patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 18 years or older
* Diabetes Mellitus (Type 1 or Type 2) undergoing treatment
* Angiographically confirmed stenosis (≥ 70%) lesion of the proximal LAD (segment 6) or mid LAD (segment 7), with no culprit lesion or stenosis of more than 60% (in a vessel of 1.5 mm or more) in the LCX and RCA territories, and no stenosis equal or more than 50% in the left main artery. Diagonal disease does not constitute an exclusion
* Angiographic characteristics amenable to both PCI/DES and MICS CABG
* Indication for revascularization based upon symptoms of angina and/or objective evidence of myocardial ischemia
* Willing to comply with all follow-up required study visits
* Signed and received copy of informed consent

Exclusion Criteria:

* Severe congestive heart failure (class III or IV according to NYHA, or pulmonary edema) at the time of enrollment.
* Left ventricular ejection fraction less than 20%;
* Prior CABG surgery.
* Prior Valve surgery.
* Prior PCI with stent implantation within 6 months.
* Previous tuberculosis or trauma to the chest that may have cause adhesions or LITA damage.
* Previous stroke within 6 months or patients with stroke at more than 6 months with significant residual neurologic involvement, as reflected in a Rankin Score > 1.
* Prior history of significant bleeding (within the previous 6 months) that might be expected to occur during CABG or PCI/DES related anticoagulation.
* In-stent restenosis in the LAD.
* Left main stenosis (50% or more).
* STEMI or Q-wave MI within 72 hours prior to enrollment
* Planned simultaneous surgical procedure unrelated to coronary revascularization (e.g. valve repair/replacement, aneurysmectomy, carotid endarterectomy or carotid stent).
* Contraindication to either CABG or PCI/DES because of a coexisting clinical condition.
* Significant leukopenia, neutropenia, thrombocytopenia, anemia, or known bleeding diathesis.
* Intolerance or contraindication to aspirin or both clopidogrel and ticagrelor.
* Dementia with a Mini Mental Status Examination (MMSE) score of <20.
* Extra-cardiac illness that is expected to limit survival to less than 5 years.
* Suspected pregnancy. A pregnancy test (urine or serum) will be administered pre-randomization to all women not clearly menopausal.
* Concurrent enrollment in another clinical trial.
* Geographically inaccessible for follow-up visits required by protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-10-01 (Estimated)

PRIMARY OUTCOMES:
Successfully enrolled, eligible and consenting patients within the first year of enrollment. | 1 year
  To determine the feasibility of the study by successfully recruiting 100 patients within the 1 year recruitment period.

SECONDARY OUTCOMES:
All-cause Mortality | 2 years
  All-cause mortality will be compared for the therapy comparison PCI/DES versus MICS CABG. For these analyses, the survival analysis outlined for the primary analysis will be followed.
Myocardial Infarction (MI) | 2 years
  MI will be compared for the therapy comparison PCI/DES versus MICS CABG. For these analyses, the survival analysis outlined for the primary analysis will be followed.
Stroke | 2 years
  Stroke will be compared for the therapy comparison PCI/DES versus MICS CABG. For these analyses, the survival analysis outlined for the primary analysis will be followed.
Target Vessel Revasularization (TVR) | 2 years
  TVR will be compared for the therapy comparison PCI/DES versus MICS CABG. For these analyses, the survival analysis outlined for the primary analysis will be followed.
Quality of Life (QOL) | 2 years
  QOL at 1 month, 6 months, 1 year, 18 months, and 2 year will be compared for the therapy comparison PCI/DES vs. MICS CABG. Patients will undergo the following QOL questionnaires at each time point above: The EuroQOL (EQ-5D), Seattle Angina Questionnaire, (SAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Ruel, MD, Principal Investigator — Ottawa Heart Institute Research Corporation

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared with other researchers/institutions unless a contract or agreement is determined.